CLINICAL TRIAL: NCT05235347
Title: Sotrovimab Expanded Access Treatment Protocol
Brief Title: Sotrovimab Expanded Access Treatment Protocol (COVID-19)
Status: No longer available | Type: Expanded Access
Sponsor: Vir Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VIR-7831-6406
Record Dates: First submitted 2022-01-13; First posted 2022-02-11 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Covid19
Keywords: SARS-CoV-2; coronavirus; coronavirus disease 2019; COVID-19
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — sotrovimab

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Biological: Sotrovimab — 500mg IV

SUMMARY:
An expanded access program for sotrovimab administered intravenously to participants with COVID-19 illness who meet current authorized/approved criteria for use of sotrovimab.

ELIGIBILITY:
Inclusion Criteria:

* In the opinion of the investigator, meets the current Emergency Use Authorization (EUA) eligibility criteria for sotrovimab

OR

* patients currently hospitalized for a non-COVID-19 illness who acquire COVID-19 (nosocomial infection) and otherwise meets all the current EUA eligibility criteria

Exclusion Criteria:

* Hospitalized due to COVID-19 (excludes nosocomial infection)
* Require oxygen therapy due to COVID-19, OR who require an increase in baseline oxygen flow rate due to COVID-19

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Site, Palo Alto, California
  - Site, Boston, Massachusetts
  - Site, St Louis, Missouri
  - Site, Seattle, Washington